CLINICAL TRIAL: NCT02183844
Title: Implementing Patient-Centered Decision Support for Mental Health
Brief Title: A System for Preference Assessment in Mental Health
Acronym: SPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government); Los Angeles County Department of Mental Health (Unknown)
Responsible Party: Principal Investigator, Alexander S. Young, MD MSHS, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R21MH100565 (NIH)
Record Dates: First submitted 2014-06-30; First posted 2014-07-08 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Mental Disorders; Schizophrenia; Overweight; Obesity
Keywords: Medical Informatics; Patient-Centered; Healthcare Preferences; Health Education; Quality Improvement; Weight Loss; Personal Satisfaction; Humans; Cognition; Body Weight
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Overweight; Obesity; Health Education; Weight Loss; Personal Satisfaction; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychosocial Weight Intervention (Experimental): Weekly group intervention for diet and exercise, designed specifically for individuals with serious mental illness and the cognitive deficits that accompany those illnesses
  Interventions: Behavioral: Psychosocial Weight Intervention

INTERVENTIONS:
Behavioral: Psychosocial Weight Intervention — Weekly group intervention for diet and exercise, designed specifically for individuals with serious mental illness and the cognitive deficits that accompany those illnesses

SUMMARY:
It is important that individuals with serious mental illness make informed choices among alternative healthcare treatments based on their preferences. However, at present, individuals' preferences are often not being elicited, nor used to guide which treatments are made available. In this pilot project, the investigators implement and evaluate a computerized method for assessing treatment preferences of individuals with schizophrenia. The investigators use weight management treatments for this initial test of the system. If this assessment method is found to predict treatment use and satisfaction, it can be used to guide implementation of treatments that improve outcomes while meeting individuals' preferences.

DETAILED DESCRIPTION:
Background/Rationale: It is important that individuals with serious mental illness have access to treatments that meet their preferences, and that they make informed choices among alternative treatments. Too often, preferences are not being routinely elicited, nor used to guide which treatments are made available. Schizophrenia is a serious mental illness that is common and produces substantial disability when poorly treated. National treatment guidelines specify that individuals with schizophrenia should receive evidence-based treatments that improve outcomes. For example, obesity is a pressing problem in this population, a side-effect of commonly used medications, and a cause of cardiovascular disease and premature mortality. There are multiple, different psychosocial interventions for weight management that can lead to reduced weight. None are widely used. If individuals' preferences were routinely assessed, then clinicians and managers would know when to make alternative treatments available.

Objectives: This project implements and evaluates a method for routinely assessing the treatment preferences of individuals with schizophrenia. The objectives are to: 1) develop a computerized, kiosk-based system that delivers education regarding treatment options for weight, uses conjoint analysis to elicit preferences, and meets the cognitive needs of individuals with schizophrenia; 2) study the feasibility and acceptability of implementing this method at a mental health clinic; and, 3) evaluate the extent to which this method predicts use of evidence-based weight services, and satisfaction with services at three months.

Methods: This is a prospective evaluation of preferences, treatment use, and satisfaction in individuals with schizophrenia. 94 individuals are enrolled who are overweight and receiving treatment at a busy, urban mental health clinic. These participants use a kiosk system that provides them with education about treatment options, and assesses their preferences regarding alternative treatments for weight. They are then offered a weekly, intensive, evidence-based psychosocial treatment for weight. Research assessments occur at baseline and 3 months. Treatment preferences are analyzed to determine how they relate to use of weight treatment, and satisfaction with treatment.

Significance: People with serious mental illness could benefit from access to effective treatments. Implementing these treatments would be facilitated by routinely collecting information regarding individuals' preferences. If the assessment method in this study is found to be feasible, acceptable, and accurate, it could be used to support implementation of improved care at clinics, medical centers, and community-based programs.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of schizophrenia
2. age 18 or older
3. Body Mass Index (BMI) of either 28.0-29.9 and gained 10 pounds in the last 3 months; OR, BMI of 30 or above
4. able to provide informed consent

Exclusion Criteria:

1. a medical condition for which a weight program is contraindicated
2. pregnant and nursing mothers
3. attendance at a psychosocial intervention for weight management in the past month
4. individuals with legal conservators who manage informed consent
5. can not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Days until using weight services | 3 months
  Utilization of the weight services offered. This includes the number of days until starting to use weight services. This is assessed using information regarding attendance at weight services, and by survey administered by interview.
Participant preferences regarding weight services | Baseline
  Individuals' preferences are assessed regarding different attributes of weight treatments. These are assessed using computerized conjoint analysis methods.
Satisfaction with the weight services provided | 3 months
  Satisfaction with the weight services provided. This is assessed using the Client Satisfaction Questionnaire administered by interview.
Number of weight services used | 3 months
  Utilization of the weight services offered. This includes the number of weight service sessions attended. This is assessed using information regarding attendance at weight services, and by survey administered by interview.

SECONDARY OUTCOMES:
Feasibility and acceptability of implementing preference assessment | Baseline
  Feasibility and acceptability of implementing kiosk-based preference assessment at a mental health clinic. This is assessed using project records, surveys, and semi-structured interview questions assessing whether participants and staff find the program and its components to be advantageous, relevant, simple, easy to use, and beneficial.

OTHER OUTCOMES:
Aspects of the Theory of Planned Behavior | Baseline and 3 months
  Attitudes, subjective norms, perceived control, and behavioral intentions regarding weight loss. These are assessed by interview, using scales from the Theory of Planned Behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Young, MD, MSHS, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Health Services and Society, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young AS, Niv N, Chinman M, Dixon L, Eisen SV, Fischer EP, Smith J, Valenstein M, Marder SR, Owen RR. Routine outcomes monitoring to support improving care for schizophrenia: report from the VA Mental Health QUERI. Community Ment Health J. 2011 Apr;47(2):123-35. doi: 10.1007/s10597-010-9328-y. Epub 2010 Jul 25. PMID 20658320
- [Background] Cohen AN, Chinman MJ, Hamilton AB, Whelan F, Young AS. Using patient-facing kiosks to support quality improvement at mental health clinics. Med Care. 2013 Mar;51(3 Suppl 1):S13-20. doi: 10.1097/MLR.0b013e31827da859. PMID 23407006
- [Background] Brown AH, Cohen AN, Chinman MJ, Kessler C, Young AS. EQUIP: implementing chronic care principles and applying formative evaluation methods to improve care for schizophrenia: QUERI Series. Implement Sci. 2008 Feb 15;3:9. doi: 10.1186/1748-5908-3-9. PMID 18279505
- [Background] Chinman M, Young AS, Schell T, Hassell J, Mintz J. Computer-assisted self-assessment in persons with severe mental illness. J Clin Psychiatry. 2004 Oct;65(10):1343-51. doi: 10.4088/jcp.v65n1008. PMID 15491237
- [Background] Young AS. The client, the clinician, and the computer. Psychiatr Serv. 2010 Jul;61(7):643. doi: 10.1176/ps.2010.61.7.643. No abstract available. PMID 20591993